CLINICAL TRIAL: NCT05847400
Title: Predictors of Chronic Kidney Disease Among Type 2 Diabetic Patients in Assiut University Hospitals
Acronym: Ckd&dm
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Muhammed Ali Aboalsaud, Aboalsaud, Assiut University
Other Study IDs: ckd in tybe 2 dm
Record Dates: First submitted 2023-04-27; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Type 2 Diabetes With Renal Manifestations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CKD patients with T2DM on regular HD: CKD patients with T2DM attending Assuit university diabetic outpatients clinic and ESRD on regular HD at dialysis unit of Assuit University Hospital
- CKD patients with T2DM not on regular HD: CKD patients with T2DM attending Assuit university diabetic outpatients clinic and ESRD not on regular HD at dialysis unit of Assuit University Hospital

SUMMARY:
Predictors of Chronic Kidney Disease among Type 2 Diabetic Patients in Assiut University Hospitals.

DETAILED DESCRIPTION:
Globally, the total number of people with diabetes is estimated to increase from 415 million (8.8%) in 2015 to 642 million (10.4%) in 2040, with the largest alterations expected to occur in the urban population of low- to middle-income countries (LMICs)1. Of them, type 2 diabetes mellitus (T2DM) accounts for more than 90% of people with diabetes2,3. By 2040, the difference worldwide is projected to broaden, with 477.9 million affected people living in urban areas and 163.9 million in rural areas1. It has been postulated that the burden of diabetes and its complications in the LMICs may be contributed by the economic development and rapid urbanisation via increased caloric intake and the adoption of a sedentary lifestyle2,4,5. More importantly, the most striking demo graphic change to diabetes prevalence in global terms also seems to be related to the growth of the proportion of the elderly population6. Despite rates of diabetes-related complications such as CVDs decreasing significantly in the past two decades, it has not translated nearly as well as kidney complications7. Approximately 10% of deaths in people with T2DM are attributable to kidney failure8. It is well-established that diabetes-related chronic kidney disease (CKD) is the leading cause of end-stage kidney disease (ESKD) in T2DM patients worldwide9,10.

In our study, we aim to identify and classify patients attending diabetic outpatient clinic with both CKD and

ELIGIBILITY:
Inclusion Criteria:

- Patients with T2DM aged 18 years or older. For patients whom eGFR values < or =60 ml/min/1.73m2.

Patient with type 2 DM and ESRD on regular HD with duration less than 1 year

Exclusion Criteria:

Having kidney transplantation incomplete data on glycemic control. Patients with type 2 DM and ESRD on regular HD with duration more than 1 year. Pregnant woman. Patients with advanced comorbides(cardiac, hepatic,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All type 2 diabetic &ckd patient older than 18 years
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-03-28 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
predictors of CKD among T2DM patients attending Assiut University Hospitals. To classify our patients into stages according to KDIGO guidelines | 3 years
  To identify predictors of CKD among T2DM patients attending Assiut University Hospitals.
  To classify our patients into stages according to KDIGO guidelines

SECONDARY OUTCOMES:
the possible risk factors contributing to progessing CKD in T2DM patients. | 3 years
  To identify the possible risk factors contributing to progessing CKD in T2DM patients.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammed Al Abualsaud, Principal Investigator — Assiut University
Locations (1):
- Assiut, Asyut, Egypt